CLINICAL TRIAL: NCT01630850
Title: Islet Transplantation in Patients With "Brittle" Type I Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0684
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogenic islet cells (human, U. Chicago) (Experimental)
  Interventions: Biological: Allogenic islet cells (human, U. Chicago); Procedure: Intraportal infusion of islet cells

INTERVENTIONS:
Biological: Allogenic islet cells (human, U. Chicago) — Human allogenic islet cells. Immunosuppression may include remicade, thymoglobulin,prograf, solu-medrol, and cellcept. Dosage will vary per patient based on weight. Patients will receive immunosuppression medications while islet cells are functioning.
Procedure: Intraportal infusion of islet cells — Intraportal infusion of islet cell through the portal vein in the liver.

SUMMARY:
The purpose of this study is to learn about the safety of islet transplantation for Type 1 diabetes mellitus, which may provide more normal control of blood sugar without the need for insulin shots. Islets are special clusters of cells within the pancreas that produce insulin. These cells will be obtained from cadaver (non-living) donors and given to subjects by vein.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 70 years of age.
* Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
* Clinical history compatible with T1D with onset of disease at < 40 years of age, insulin-dependence for ≥ 5 years at the time of enrollment, and a sum of patient age and insulin dependent diabetes duration of ≥ 28 and absent stimulated c-peptide (<0.3ng/mL) in response to a mixed meal tolerance test (MMTT; Boost® 6 mL/kg body weight to a maximum of 360 mL; another product with equivalent caloric and nutrient content may be substituted for Boost) measured at 60 and 90 min after the start of consumption and at least one episode of severe hypoglycemia in the 12 months prior to study enrollment; OR a clinical history of "problematic hypoglycemia" defined as defined as two or more episodes per year of severe hypoglycemia or as one episode associated with impaired awareness of hypoglycemia, extreme glycemic lability, or major fear and maladaptive behavior according to recent clinical recommendations.
* Involvement in intensive diabetes management defined as self monitoring of glucose values no less than a mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy. Such management must be under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least 3 clinical evaluations during the 12 months prior to study enrollment.
* Reduced awareness of hypoglycemia as defined by a Clarke score of 4 or more OR a HYPO score greater than or equal to the 90th percentile (1047) during the screening period and within the last 6 months; OR marked glycemic lability characterized by wide swings in blood glucose despite optimal diabetes therapy and defined by an LI score greater than or equal to the 90th percentile (433 mmol/L2/h -wk1) during the screening period and within the last 6 months prior to randomization; OR a composite of a Clarke score of 4 or more and a HYPO score greater than or equal to the 75th percentile (423) and a LI greater than or equal to the 75th percentile (329) during the screening period and within the last 6 months.

Exclusion Criteria:

* Body mass index (BMI) >30 kg/m2 or patient weight <50kg.
* Insulin requirement >1.0 IU/kg/day or <15 U/day.
* Untreated proliferative diabetic retinopathy.
* Blood Pressure: SBP >160 mmHg or DBP >100 mmHg.
* Measured glomerular filtration rate <80 mL/min/1.73m2 (using iohexol or calculated using the subject's measured serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI equation) or based on 24-hrs urine collection. Strict vegetarians (vegans) with a calculated GFR <70 mL/min/1.73m2 are excluded. The absolute (raw) GFR value will be used for subjects with body surface areas >1.73 m2.
* Presence or history of macroalbuminuria (>300 mg/g creatinine).
* Presence or history of panel-reactive anti-HLA antibodies above 30% or history/presence of donor specific anti-HLA antibodies in order to avoid unacceptable antigen(s) (Campbell PM 2007).
* For female subjects: Positive pregnancy test, presently breast-feeding, wishes to be pregnant at any time point in the future, which includes during or after the completion of the study even if study participation is ended early, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.
* Known active alcohol or substance abuse.
* Severe co-existing cardiac disease
* Known hypercoagulative state.
* Symptomatic cholecystolithiasis.
* Acute or chronic pancreatitis.

Other protocol related inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
HbAlc <7.0% and an absence of severe hypoglycemic events | 1 year
  The proportion of subjects with an HbAlc <7.0% at Day 365 AND free of severe hypoglycemic events from Day 28 to Day 365 inclusive following the first islet transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Witkowski, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Wang Q, Huang YX, Liu L, Zhao XH, Sun Y, Mao X, Li SW. Pancreatic islet transplantation: current advances and challenges. Front Immunol. 2024 Jun 3;15:1391504. doi: 10.3389/fimmu.2024.1391504. eCollection 2024. PMID 38887292
- [Background] Lee J, Yoon KH. Islet transplantation in Korea. J Diabetes Investig. 2024 Sep;15(9):1165-1170. doi: 10.1111/jdi.14264. Epub 2024 Aug 6. PMID 39105663
- [Background] Spence KT, Ladie DE. Islets Transplantation. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK562272/ PMID 32965943
- [Background] Wang S, Du Y, Zhang B, Meng G, Liu Z, Liew SY, Liang R, Zhang Z, Cai X, Wu S, Gao W, Zhuang D, Zou J, Huang H, Wang M, Wang X, Wang X, Liang T, Liu T, Gu J, Liu N, Wei Y, Ding X, Pu Y, Zhan Y, Luo Y, Sun P, Xie S, Yang J, Weng Y, Zhou C, Wang Z, Wang S, Deng H, Shen Z. Transplantation of chemically induced pluripotent stem-cell-derived islets under abdominal anterior rectus sheath in a type 1 diabetes patient. Cell. 2024 Oct 31;187(22):6152-6164.e18. doi: 10.1016/j.cell.2024.09.004. Epub 2024 Sep 25. PMID 39326417
- [Background] Ghoneim MA, Gabr MM, El-Halawani SM, Refaie AF. Current status of stem cell therapy for type 1 diabetes: a critique and a prospective consideration. Stem Cell Res Ther. 2024 Jan 29;15(1):23. doi: 10.1186/s13287-024-03636-0. PMID 38281991
- [Background] El Nahas R, Al-Aghbar MA, Herrero L, van Panhuys N, Espino-Guarch M. Applications of Genome-Editing Technologies for Type 1 Diabetes. Int J Mol Sci. 2023 Dec 26;25(1):344. doi: 10.3390/ijms25010344. PMID 38203514